CLINICAL TRIAL: NCT01812902
Title: Prospective Randomized Study Comparing Extended With Limited Pelvic Lymphadenectomy in Intermediate and High Risk Prostate Cancer Patients Undergoing Radical Prostatectomy
Brief Title: Prospective Study Comparing Extended With Limited Pelvic Lymphadenectomy in Intermediate and High Risk Prostate Cancer Patients Undergoing Radical Prostatectomy
Acronym: LFD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Marcos Francisco Dall'Oglio, M.D. Phd, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UROUSP - 006
Record Dates: First submitted 2013-03-12; First posted 2013-03-18 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Prostate specific antigen; lymphadenectomy; Limited lymphadenectomy; Extended lymphadenectomy; Immunohistochemistry
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extended LND (Experimental): Radical Prostatectomy with extended lymphadenectomy
  Interventions: Procedure: Radical Prostatectomy
- Limited LND (Active Comparator): Radical Prostatectomy with Limited lymphadenectomy
  Interventions: Procedure: Radical Prostatectomy

INTERVENTIONS:
Procedure: Radical Prostatectomy

SUMMARY:
Prostate cancer is currently the second most common cause of cancer death in men in Western countries. Lymphadenectomy is the gold standard procedure for staging pelvic lymph node and is classically indicated in intermediate and high risk prostate cancer patients and is held at the same time of prostatectomy. A traditionally pelvic lymphadenectomy covers the obturator chain bilaterally. Recently, some studies have demonstrated the existence of lymph node involvement outside the traditional boundaries of classical lymphadenectomy, recommending therefore extended dissection; this also includes the external / internal / common iliac chains and presacral. Thus lymphadenectomy, according to these authors, would also has a therapeutic role, besides helping in better staging. Although some retrospective studies report an association between lymphadenectomy and tumor progression, the exact impact of extended lymphadenectomy in oncological outcome of patients with prostate cancer is not clearly established, mainly by lack of prospective randomized studies on the subject . The study objectives are to compare the oncologic results of extended lymphadenectomy versus limited in order to elucidate the role of extended dissection in lymph node staging and results of treatment in terms of increased tumor cure. The investigators also intend to identify patients who may benefit from oncologically extended procedure. To do this, the investigators will evaluate prospectively patients diagnosed with prostate cancer at intermediate or high risk indicating lymphadenectomy and radical prostatectomy. These patients will be randomized to the extended versus limited lymphadenectomy and the investigators will compare the lymph node metastasis and pattern of spread of prostate cancer, as well as biochemical relapse-free survival, freedom from progression to metastasis and cancer-specific survival.

ELIGIBILITY:
Inclusion Criteria:

* Prostate Cancer patients with intermediate or high risk and with indication of radical prostatectomy and LND
* Absence of bone metastasis or other organ imaging test (MRI or scintigraphy)
* Absence of hormone treatment
* Absence of radiotherapy
* Signing an informed consent
* Availability and adequacy of lymph node tissue samples to perform the immunohistochemical

Exclusion Criteria:

* Life expectancy less than 10 years
* Absence of clinical conditions for the procedure
* Laparoscopic or perineal surgery
* Presence of bone or visceral metastasis
* Neoadjuvant treatment
* Another malignant neoplasia
* Prior abdominal or pelvic surgery

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2012-02; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Biochemical relapse-free survival | Five years

SECONDARY OUTCOMES:
Staging | One Month
  At the moment of the pathological analysis We will do immunohistochemistry to detect micro metastasis
Cancer specific survival | 10 years

OTHER OUTCOMES:
Spread pattern of prostate cancer | One Month
Metastasis free survival | Ten years

CONTACTS AND LOCATIONS:
Overall Officials: Marcos F Dall'Oglio, M.D. Phd, Study Director — University of Sao Paulo; Jean FP Lestingi, Doctor, Principal Investigator — University of Sao Paulo; Jose P Junior, M.D, Study Chair — University of Sao Paulo; Alexandre C Sant'Anna, M.D, Study Chair — University of Sao Paulo; Rafael F Coelho, Doctor, Study Chair — University of Sao Paulo; Giuliano B Guglielmetti, Doctor, Study Chair — University of Sao Paulo; Juliana N Ravaninni, Doctor, Study Chair — University of Sao Paulo; Daher C Chade, M.D., Study Chair — University of Sao Paulo; Matheus S Chaib, Doctor, Study Chair — University of Sao Paulo; Mauricio D Cordeiro, Doctor, Study Chair — University of Sao Paulo; Rodrigo R Pessoa, Doctor, Study Chair — University of Sao Paulo; Luiz AA Botelho, Doctor, Study Chair — University of Sao Paulo; Adriano Nesralla, M.D., Study Chair — University of Sao Paulo; Claudio B Murta, Doctor, Study Chair — University of Sao Paulo; Fabio L Ortega, Doctor, Study Chair — University of Sao Paulo; Daniel K Abe, M.D., Study Chair — University of Sao Paulo; Leonardo L Borges, Doctor, Study Chair — University of Sao Paulo; Luiz CN Oliveira, M.D., Study Chair — University of Sao Paulo; Flavio GM Areas, Doctor, Study Chair — University of Sao Paulo
Locations (1):
- Instituto do Cancer do Estado de São Paulo, São Paulo, Brazil